CLINICAL TRIAL: NCT07392905
Title: Association Between Food Intake-Related Brain Functional Patterns and Metabolic Profiles in Patients With Obesity: A Randomized Crossover Trial
Brief Title: Food Intake-Related Brain and Metabolic Responses in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-0875-02
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Brain Function; Metabolomics; Feeding Behavior; Macronutrients
Keywords: obesity; macronutrient; fMRI; Cross-over trial; Plasma metabolome; Satiety; Nutrient challenge
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose Challenge (Experimental): Participants receive a single 200 kcal liquid meal consisting of 50 g glucose powder dissolved in water to a final volume of 300 mL, administered 6 hours after consuming a standardized pre-load meal.
  Interventions: Dietary Supplement: Glucose Liquid Meal
- Fat Challenge (Experimental): Participants receive a single 200 kcal liquid meal consisting of 100 mL intralipid emulsion diluted with water to a final volume of 300 mL, administered 6 hours after consuming a standardized pre-load meal.
  Interventions: Dietary Supplement: Fat Liquid Meal
- Protein Challenge (Experimental): Participants receive a single 200 kcal liquid meal consisting of 54 g whey protein isolate powder dissolved in water to a final volume of 300 mL, administered 6 hours after consuming a standardized pre-load meal.
  Interventions: Dietary Supplement: Protein Liquid Meal

INTERVENTIONS:
Dietary Supplement: Glucose Liquid Meal — A standardized, isocaloric (200 kcal), isovolumetric (300 mL) liquid meal containing 50 g pure glucose. Administered orally 6 hours after a standardized pre-load meal.
  Arms: Glucose Challenge
Dietary Supplement: Fat Liquid Meal — A standardized, isocaloric (200 kcal), isovolumetric (300 mL) liquid meal prepared from 100 mL of intralipid emulsion diluted with water. Administered orally 6 hours after a standardized pre-load meal.
  Arms: Fat Challenge
Dietary Supplement: Protein Liquid Meal — A standardized, isocaloric (200 kcal), isovolumetric (300 mL) liquid meal containing 54 g whey protein isolate powder. Administered orally 6 hours after a standardized pre-load meal.
  Arms: Protein Challenge

SUMMARY:
This study is a prospective, single-center, randomized, controlled, crossover intervention trial. A total of 60 participants, including 30 patients with obesity and 30 healthy controls, will be enrolled. Each participant will receive an isocaloric liquid meal challenge (glucose, fat, or protein) on three separate experimental days, with a washout period of at least 7 days between visits to eliminate carryover effects from the previous intervention. The primary objective is to investigate the association between brain functional patterns and plasma metabolic profiles following the ingestion of different macronutrients in patients with obesity, aiming to uncover potential neuro-metabolic imbalance features.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized, controlled, crossover intervention trial enrolling 60 participants, including 30 obese patients and 30 healthy control volunteers. Each participant will be randomly assigned to one of the six possible sequences of three macronutrient interventions (A: glucose, B: fat, C: protein)-namely ABC, ACB, BAC, BCA, CAB, or CBA-to ensure balanced allocation across intervention orders. Each participant will undergo one nutrient challenge on each of three separate experimental days, with at least a 7-day washout period between visits to minimize carryover effects from prior interventions. During the washout periods, participants are required to maintain stable habitual dietary patterns and avoid extreme diets, high-intensity exercise, irregular sleep schedules, and intake of additional nutritional supplements; adherence will be monitored via brief diet and activity logs.

The intervention consists of isocaloric (200 kcal) and isovolumetric (300 mL) liquid meals, specifically formulated as follows: Glucose arm: 50 g glucose powder dissolved in water to a final volume of 300 mL; Fat arm: 100 mL intralipid emulsion diluted with water to a final volume of 300 mL; Protein arm: 54 g whey protein powder dissolved in water to a final volume of 300 mL. On each experimental day, participants must arrive in a fasting state. Prior to nutrient administration, they will complete clinical laboratory tests, body composition assessment, hepatic fat quantification, and eating behavior questionnaires. During and after the intervention, participants will provide dynamic postprandial satiety ratings, multi-timepoint blood and stool samples (for untargeted metabolomic analysis), and undergo functional magnetic resonance imaging (fMRI) within a predefined postprandial time window. Finally, neuroimaging metrics, peripheral metabolomic profiles, and subjective satiety scores will be integrated through multidimensional correlation analyses to explore the neuro-metabolic coupling responses to different macronutrient challenges in obesity, thereby providing theoretical insights and potential targets for precision nutrition interventions.

ELIGIBILITY:
Inclusion Criteria:

Obese participants:

1. BMI ≥ 28 kg/m²;
2. Age 18-40 years;
3. Any gender;
4. Right-handed.

Healthy control participants:

1. BMI 18.5-23.9 kg/m²;
2. Age 18-40 years;
3. Any gender;
4. Right-handed.

Exclusion Criteria:

1. Diabetes mellitus;
2. Contraindications or allergies to any ingredient in the standardized meal or macronutrient challenges used in this study;
3. Central nervous system disorders (e.g., traumatic brain injury, acute cerebral infarction, epilepsy) or psychiatric disorders (e.g., depression, schizophrenia); use of medications acting on the central nervous system within the past 3 months or long-term use;
4. Severe impairment of liver, kidney, heart, or gastrointestinal function, including alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels >2 times the upper limit of normal; estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m² calculated by the CKD-EPI equation; history of unstable angina or myocardial infarction within the past 3 months, or heart failure classified as New York Heart Association (NYHA) class II or higher; history of gastrointestinal stoma, bowel resection, intestinal obstruction, or peptic ulcer disease;
5. Contraindications to MRI, such as implanted metallic devices or claustrophobia;
6. Pregnancy or lactation;
7. Participation in another clinical trial currently or within the past 3 months; use of nutritional supplements within the past 3 months or long-term use;
8. History of prior metabolic/bariatric surgery;
9. Use of antibiotics or probiotics within the past 1 month;
10. Use of medications affecting metabolism or causing weight loss within the past 1 month; body weight fluctuation exceeding 3 kg during the month prior to screening;
11. Unusual dietary habits; daily alcohol intake >40 grams, smoking >10 cigarettes per day, or coffee consumption ≥2 cups per day.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-21 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Acute Brain Functional Response to Macronutrient Challenges | Baseline (pre-challenge) and within 0-20 minutes post-challenge on each experimental day
  Changes in whole-brain functional activation patterns assessed by blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (fMRI), comparing pre-challenge baseline with post-challenge scans acquired within 20 minutes after ingestion of glucose, fat, or protein.
Dynamic Plasma Metabolomic Response to Macronutrient Challenges | Baseline (pre-challenge), 30 minutes post-challenge, and 120 minutes post-challenge on each experimental day.
  Temporal changes in plasma metabolic profiles characterized by untargeted metabolomic profiling, evaluating the evolution of metabolite concentrations across three time points: before intervention, 30 minutes post-intervention, and 120 minutes post-intervention, following single-dose challenges with glucose, fat, or protein.

SECONDARY OUTCOMES:
Temporal Changes in Subjective Satiety and Hunger Ratings | Pre-challenge, 0 minutes, 30 minutes, and 120 minutes post-challenge on each experimental day.
  Subjective levels of satiety and hunger assessed using a standardized visual analog scale (VAS), with ratings collected at four time points: before nutrient challenge, immediately after ingestion (0 minutes), 30 minutes post-challenge, and 120 minutes post-challenge.
Inter-group Differences in Brain Functional and Metabolic Responses Between Obese and Healthy Participants | Baseline, within 0-20 minutes (fMRI), and 30/120 minutes (metabolomics) post-challenge on each experimental day
  Comparison of whole-brain fMRI activation patterns and plasma metabolomic profiles between obese participants and healthy controls following glucose, fat, or protein challenges, to evaluate group-level differences in neuro-metabolic responsiveness.
Changes in Gut Microbiota Composition and Alpha/Beta Diversity Following Macronutrient Challenges | Approximately 24 hours before intervention and approximately 24 hours after intervention on each experimental day
  Fecal samples collected approximately 24 hours before and 24 hours after each macronutrient challenge are analyzed via 16S rRNA gene sequencing (or metagenomic sequencing) to assess changes in gut microbial composition, alpha diversity (within-sample), and beta diversity (between-sample).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, Principal Investigator — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Department of Endocrinology, Endocrine and Metabolic Disease Medical Center,Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No